CLINICAL TRIAL: NCT00886756
Title: A Phase I, Single-Centre, Randomised, Double-Blind, Placebo Controlled Single-Ascending Dose, Study to Assess the Safety, Tolerability, Pharmacokinetics of AZD8529 in Healthy Male Japanese Subjects
Brief Title: AZD8529 Single Ascending Dose Study in Healthy Japanese Subjects
Acronym: JSAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1960C00003; 2009-009940-22
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Phase I; Japanese healthy volunteer; AZD8529
MeSH Terms: interventions — AZD8529

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8529
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8529 — Oral
  Arms: 1
Drug: Placebo — Oral
  Arms: 2

SUMMARY:
This is a Phase I, double-blind, placebo-controlled, randomised within each dose group, single ascending dose study, with the objective to assess the safety, tolerability and pharmacokinetic profile of AZD8529 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese subjects aged 20 to 45 years (inclusive)
* Have a body mass index (BMI) between 18 and 27 kg/m 2 (inclusive) and weigh at least 50 kg.least 50 kg.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Any clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, haematology or urinalysis as judged by the Investigator and/or Sponsor.
* Smoking in excess of 5 cigarettes per day or the equivalent within 28 days of Day 1.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-04; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To asses the safety:Adverse events, vital signs, physical examinations, telemetry, dECGs, clinical chemistry and haematology labs including testosterone, prolactin, LH, FSH and TSH, and urinalysis. | From screening period to follow-up, 42 days (maiximum).

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD8529 in plasma and urine. | Blood and urine sampling from pre-dose until 12 days post dose.
To collect and store DNA for future exploratory research | One blood sampling after randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD MFPM FRCA, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Research Site, London, United Kingdom